# Official Title of the study: Effects of Intermittent Fasting in Metabolic Dysfunction Associated Fatty Liver Disease

NCT number: NCT06664684

Date of the document: 06.05.2022

### Study Protocol

#### **Patients**

This study was approved by the Ethics Committee of Marmara University School of Medicine (No: 09.2022.707) Informed consent was obtained from each patient included in the study. This is a prospective non-drug intervention study conducted by the same gastroenterologist on patients diagnosed with MAFLD. Individuals with fatty liver disease diagnosed by vibration-controlled transient elastography are diagnosed with MAFLD if at least one of the following three conditions is present: overweight/obesity, type 2 diabetes mellitus (T2DM), or underweight or normal weight with at least two metabolic risk abnormalities [waist circumference, blood pressure, triglycerides, high-density lipoprotein cholesterol (HDL-C), prediabetes, insulin resistance, high-sensitivity C reactive protein (CRP)]. All of our patients were diagnosed with MAFLD because their BMI was above 25 kg/m2 in addition to the detection of fatty liver.

Exclusion criteria were patients with an average daily alcohol consumption of >20 g for females and >30 g for males; pregnant or lactating women; patients with ischemic heart disease or heart failure, chronic inflammatory diseases, chronic viral infections, cancer, moderate-to-severe kidney disease, uncontrolled hypertension, and eating disorders; those with a history of bariatric surgery; and those on insulin due to increased risk of hypoglycemia.

#### Design

Patients who voluntarily agreed to participate in the study were randomly assigned into two groups. Patients enrolled in the study were referred for an initial consultation with a dietitian following their diagnosis by a gastroenterologist. The energy-restricted diet group followed an energy-restricted diet for 8 weeks, while the energy + time-restricted diet group followed the same diet and a 16:8 eating pattern and restricted food intake to an 8 h window each day. The effectiveness of the intervention was assessed using anthropometric and biochemical measurements, and Fibroscan investigations were performed before the intervention (T0) and after the intervention (T8).

## Measurements

Blood samples were collected from patients after 12 h of fasting. The samples were centrifuged for 15 min and stored at –80 °C after serum separation until analysis. Serum FGF-21, Beclin-1, and ATG-5 were analyzed using enzyme-linked

immunosorbent assay (ELISA) kits, following the manufacturer's protocols (Human FGF-21 ELISA, Biovendor, Brno, Czech Republic; Human BECN1 [Beclin-1] ELISA Kit, ElabScience, Houston, TX, USA; Human Autophagy protein 5 [ATG5] ELISA Kit, MyBioSource, Inc., San Diego, USA) and in duplicate.

- The extent of hepatic steatosis and fibrosis was determined using transient elastography on a Fibroscan 502 TouchR device(Echosens SA, Paris, France). All Fibroscan measurements were performed following the manufacturer's instructions as specified previously.
- Patients' heights were measured using a stadiometer (Seca 769), barefoot, feet side by side, and head in the Frankfort plane. Body composition was determined using the bioelectrical impedance method (Tanita MC 780 P).

